CLINICAL TRIAL: NCT05541731
Title: Implementation Study of the ICOPE Program for the Detection of Frailty in the Elderly Within the Territorial Health Professional Communities (CPTS) of Brest Region
Acronym: ICOPE 29
Status: Terminated | Type: Observational
Why Stopped: Coordinator decision
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC22.0102
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Frailty is a geriatric syndrome resulting from a decrease in physiological reserve capacities altering the mechanisms of adaptation to stress with, in the absence of diagnosis and management, a short-term risk of falls, hospitalization, loss of autonomy and death.

In 2019, the World Health Organization has taken up this subject with the objective of reducing the number of dependent people in the world by 15 million, i.e. 150,000 in France. For this purpose, recommendations for integrated care for seniors (Integrated Care for Older People = ICOPE) have been published.

6 functions are essential to maintain autonomy: mobility, memory, sight, hearing, mental health and nutrition. The first step of the ICOPE program consists of screening for a decline in one of these functions using a tool made up of questions or tests that can be carried out in 8 to 10 minutes in primary care by trained non-professionals. The second step is a thorough evaluation of the person screened, leading to the creation of a personalized care plan. In the current state of affairs, despite its recommendations, this identification is not carried out in Brittany.

The objective of this study is to demonstrate the feasibility of implementing the first stage of the ICOPE program by seizing the opportunity of the creation in the Brest region of two Territorial Health Professional Communities (CPTS) : Brest Santé Océane and Iroise santé.

ELIGIBILITY:
Inclusion Criteria:

* Primary care staff belonging to one of the 2 CPTS (CPTS Brest Santé Océane and CPTS Iroise santé) and having accepted to participate in the study

Exclusion Criteria:

* Refusal to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All primary care staff in the two CPTS caring for non-dependent patients aged 70 and over
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Feasibility of identifying frail elderly people aged 70 and over | Month 12
  Number of patients screened using the ICOPE (Integrated Care for Older People) program by the primary care professionals of the CPTS Brest Santé Océane and Iroise santé, one in an urban environment and the other in a semi-rural environment.
  To demonstrate the feasibility of identifying frail elderly people aged 70 and over, using the ICOPE program, by health professionals working in two CPTSs, Brest Santé Océane and Iroise santé, .

SECONDARY OUTCOMES:
Rate of individuals who had one or more of the 6 essential functions for maintaining independence | Month 12
  Calculate the rate of individuals who had one or more of the 6 identified as impaired by the use of the ICOPE program in these two territories.
  Number of patients for whom one or more of the 6 functions (mobility, memory, sight, hearing, mental health and nutrition) essential for maintaining autonomy is impaired using the ICOPE MONITOR application. This developed by the Gerontopôle of the Toulouse University Hospital, allows the measurement of the capacities necessary for the prevention of dependency in a few minutes. This application can be downloaded free of charge for health professionals, on a smartphone or tablet.
  The assessment of the ICOPE MONITOR application consists of a series of 9 questions, an auditory examination (whisper test) and a chair rise test (have the patient rise from a chair with arms crossed over the chest 5 times in a row as quickly as possible). This assessment identifies whether the patient has any of the 6 impaired functions.
Feeling about the ICOPE MONITOR tool | Month 12
  Perception of the ICOPE MONITOR tool by professionals (qualitative study using semi-structured interviews and group interviews). There are no score.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Cpts Brest Sante Oceane, Guipavas
  - Cpts Pays D'Iroise, Saint-Renan

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending five years following the last visit of the last patient.
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Pellen N, Beurton-Couraud L, Goff-Coquet AL, Tramecon A, Gentric A, Le Reste JY. Five reasons for the failure of frailty screening in primary care: lessons from the experience with ICOPE monitor step 1. BMC Geriatr. 2025 Nov 26;25(1):1059. doi: 10.1186/s12877-025-06789-6. PMID 41299329